CLINICAL TRIAL: NCT04154449
Title: Effect of Intranasal Insulin on Postoperative Cognitive Dysfunction in Middle Aged Patients Undergoing Non Cadiac Surgery.
Brief Title: Effect of Intranasal Insulin on Postoperative Cognitive Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Nourhan mohamed anter, Resident of anesthesia and Intensive care, Minia University
Other Study IDs: 164: 2/2019
Record Dates: First submitted 2019-09-07; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Middle Aged Patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Control group.
- Surgical group Received intranasal insulin.
  Interventions: Drug: Intranasal insulin
- Surgical group Received placebo.

INTERVENTIONS:
Drug: Intranasal insulin — Surgical group Received intranasal insulin, the second group surgical Received placebo and the third group is non surgical do not receive anything.
  Groups: Surgical group Received intranasal insulin.

SUMMARY:
Our study is designed to evaluate the effect of intranasal insulin on postoperative cognitive dysfunction.

Primary outcome:

1. The occurrence of cognitive dysfunction at approximately 7 days after surgery.

Secondary outcome:

1. Incidence of any side effect.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 - 60 years.
2. Both gender.
3. Patients will be scheduled for elective major abdominal, thoracic, orthopedic, open gynecological, open urological, spine, otolaryngological surgeries under general anesthesia with expected hospital stay >4 days.

Exclusion Criteria:

* 1. Drug allergy. 2. Patients with major psychiatric disease. 3. Patients receive major tranquillizers and antidepressant. 4. Those undergoing neurosurgery or cardiac surgery. 5. Those unable or unwilling to abide by the study procedure 6. Those who could not follow procedure or who had poor comprehension of dutch language. 7. Those with sever visual and auditory disorder / handicaps.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Age 40 - 60 years.
  2. Both gender.
  3. Patients will be scheduled for elective major abdominal, thoracic, orthopedic, open gynecological, open urological, spine, otolaryngological surgeries under general anesthesia with expected hospital stay >4 days.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-12-25 (Estimated); Study Completion 2019-12-25 (Estimated)

PRIMARY OUTCOMES:
Cognitive dysfunction | 7 days
  The occurrence of cognitive dysfunction at approximately 7 days after surgery.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Minia University, Minya
  - Minia university, Minya

IPD SHARING:
Plan to Share IPD: Yes